CLINICAL TRIAL: NCT06259422
Title: Method VALIDation and Evaluation of Non-radioactive Methods to Measure Glomerular Filtration Rate
Acronym: VALIDGFR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18054
Record Dates: First submitted 2024-01-10; First posted 2024-02-14 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Kidney Function Issue; Diagnosis; Chronic Kidney Diseases
Keywords: mGFR; Kidney function; Exogenous filtration marker; Measured glomerular filtration rate; Iohexol; Iothalamate
MeSH Terms: conditions — Disease; Renal Insufficiency, Chronic | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Iohexol in addition to 125I-iothalamate and 131I-hippuran (Other): In this clinical trial, patients receiving 125I-iothalamate and 131I-hippuran during routine clinical care, will also receive iohexol. This allows us to determine the mGFR using both methods in the same patient, and compare both methods in terms of accuracy and precision.
  Interventions: Drug: Iohexol; Diagnostic Test: 125I-iothalamate and 131I-hippuran

INTERVENTIONS:
Drug: Iohexol — Subjects will receive a single bolus of 5 mL of Omnipaque 300 (containing 3235 mg iohexol)
Diagnostic Test: 125I-iothalamate and 131I-hippuran — Subjects will receive 125I-iothalamate and 131I-hippuran as part of their routine clinical care.

SUMMARY:
This study is a single centre intervention study to compare two methods of determining the measured glomerular filtration rate (mGFR). Subjects who receive radioactively labeled iothalamate (125I) and hippuran (131I) within the framework of routine clinical care, will be co-administered iohexol. The primary trial endpoint is the mGFR when administered 125I-iothalamate and 131I-hippuran versus iohexol. By determining the mGFR using both iohexol and iothalamate in the same patients, a direct comparison of the two methods can be made in terms of their accuracy and precision. This makes it possible to determine the potential use of the non-radioactive measurement method as an alternative to the radioactive method and thus lower the overall radioactive burden for patients and personnel.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a kidney function measurement test as part of standard care.
* Written informed consent.

Exclusion Criteria:

* History of hypersensitivity to iodinated contrast media or one of the excipients in the formulation of iohexol (trometamol, sodium calcium edetate, hydrochloric acid).
* Subjects with (suspected or known) thyrotoxicosis.
* Pregnant women and women of child-bearing potential who are not using reliable contraception.
* Patients who are unlikely to comply to the trial's procedure (non-compliance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
mGFR Iohexol | Through study completion, an average of 1 year
  mGFR that is determined using the iohexol method
mGFR Iothalamate and hippuran | Through study completion, an average of 1 year
  mGFR that is determined using the warm 125I-iothalamate and 131I-hippuran method

SECONDARY OUTCOMES:
Repeated mGFR using iohexol on a separate study day | Through study completion, an average of 1 year
  mGFR that is determined using the iohexol method
Repeated mGFR using iothalamate and hippuran on a separate study day | Through study completion, an average of 1 year
  mGFR that is determined using the warm 125I-iothalamate and 131I-hippuran method

OTHER OUTCOMES:
Subgroup analysis mGFR | Through study completion, an average of 1 year
  A subgroup analysis will be performed to assess whether precision and accuracy of the mGFR are dependent on important patient characteristics. This will be assessed per subgroup depending on the glomerular filtration rate (GFR) of the patients (patients with a mGFR: <30, 30-90, >90)
Subgroup analysis sex | Through study completion, an average of 1 year
  A subgroup analysis will be performed to assess whether precision and accuracy of the mGFR are dependent on the sex of the patient.
Subgroup analysis age | Through study completion, an average of 1 year
  A subgroup analysis will be performed to assess whether precision and accuracy of the mGFR are dependent on the age of the patient.
Subgroup analysis BMI | Through study completion, an average of 1 year
  A subgroup analysis will be performed to assess whether precision and accuracy of the mGFR are dependent on the BMI of the patient.
Subgroup analysis creatinine | Through study completion, an average of 1 year
  A subgroup analysis will be performed to assess whether precision and accuracy of the mGFR are dependent on the creatinine levels of the patient.
Subgroup analysis cystatin C | Through study completion, an average of 1 year
  A subgroup analysis will be performed to assess whether precision and accuracy of the mGFR are dependent on the cystatin C levels of the patient.
Subgroup analysis BSA | Through study completion, an average of 1 year
  A subgroup analysis will be performed to assess whether precision and accuracy of the mGFR are dependent on the Body Surface Area (BSA) of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided